CLINICAL TRIAL: NCT06937723
Title: Smart Monitoring Assessing Spasticity-related Health - A Prospective Multiple Sclerosis Study With Wearables
Brief Title: Smart Monitoring Assessing Spasticity-related Health
Acronym: SMASH
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Dr. med. Marc Günter Pawlitzki, Study coordinator / PI, Heinrich-Heine University, Duesseldorf
Other Study IDs: SMASH_1.0
Record Dates: First submitted 2025-03-04; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Spasticity; Smartwatch; Wearables; Digital health tools
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MS patients: Patients with Multiple Sclerosis
  Interventions: Other: Device: Smartwatch (Withings Scanwatch)

INTERVENTIONS:
Other: Device: Smartwatch (Withings Scanwatch) — All-day monitoring of patients via smartwatch

SUMMARY:
This observational study seeks to investigate the underlying of spasticity in patients with multiple sclerosis (MS) by employing multimodal monitoring techniques. By integrating digital biomarkers alongside clinical monitoring, the investigators aim to evaluate whether digital measurements are suitable for monitoring spasticity-related everyday limitations and to compare them with established clinical scores, blood analyses and questionnaires including sores on quality of life, sleep quality or activities of daily living.

DETAILED DESCRIPTION:
The symptomatic treatment of spasticity in patients with multiple sclerosis (MS) is a major challenge for both patients and healthcare providers. However, monitoring and measuring the success or failure of treatments in clinical practice remains difficult. This is mainly due to the lack of clinical scores and biomarkers that can be easily and longitudinally collected. Existing scores (such as questionnaires and the Modified Ashworth scale) are rarely used in practice. In addition, the monitoring of side effects (such as dizziness, nausea and fatigue) is difficult in routine clinical practice and often leads to premature discontinuation or switching of treatment. As a result, therapeutic options are often exhausted prematurely. Continuous monitoring with sensitive assessments could enable a better understanding of spasticity treatment.

Approximately 50 patients with moderate and severe spasticity due to MS are to be included in the study. After inclusion, follow-up examinations are carried out every 12 weeks; a total of 3 visits are planned, including the baseline examination.

The study aims to improve the understanding of spasticity symptoms and assess them in patients through multimodal clinical and longitudinal digital measurements.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to be eligible to participate in the study:

* ≥ 18 years of age
* Diagnosis of multiple sclerosis according to the McDonald criteria of 2017
* Presence of spasticity that requires medical treatment from a medical point of view
* own and use a smartphone with Android 8.1 (or higher version) or iOS 12.3 (or higher version)
* Able to operate a smartphone

Exclusion Criteria:

* Missing informed consent
* Lack of declaration of consent
* Unwillingness or inability to use the smartphone app
* Any comorbidity that leads to impaired understanding or successful completion of the study, such as (but not limited to) psychiatric comorbidities or dementia. The decision will be made at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MS and 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Wearing time of smartwatch (daily) | 180 days
Longitudinal development of activity parameter: step count | 180 days
Longitudinal development of activity parameter: approximate distance traveled (meter) | 180 days
Longitudinal development of activity parameter: duration of soft activity (seconds) defined by Withings Description: Examples for soft activity: Sleeping, Sitting quietly, Walking slowly, Typing on a computer keyboard while seated, Watching television | 180 days
Longitudinal development of activity parameter: duration of moderate activity (seconds) defined by Withings Description: Examples for moderate activity: Walking fast, Cleaning (vacuuming, washing windows, etc.), Playing doubles tennis or badminton | 180 days
Longitudinal development of activity parameter: duration of intense activity (seconds) defined by Withings Description: Examples for intense activity: Hiking, Running, Carrying heavy loads, Riding a bike, Playing football, baseball, or tennis (singles) | 180 days
Longitudinal development of activity parameter: sum of all active time (seconds) | 180 days
Longitudinal development of activity parameter: approximate calories burned Time | 180 days
Longitudinal development of sleep parameter: time awake (seconds) | 180 days
Longitudinal development of sleep parameter: number of times user woke up | 180 days
Longitudinal development of sleep parameter: time to sleep (seconds) | 180 days
Longitudinal development of sleep parameter: total time in bed (seconds) | 180 days
Longitudinal development of sleep parameter: total time asleep (seconds) | 180 days
Longitudinal development of sleep parameter: ratio of sleep/time in bed | 180 days
Longitudinal development of sleep parameter: time spent in bed before falling asleep (seconds) | 180 days
Longitudinal development of sleep parameter: time awake after first falling asleep (seconds) | 180 days
Longitudinal development of sleep parameter: Withings Sleep score Description: Defined by Withings as follows: It measures every night's sleep and provides a score out of 100 points | 180 days
Longitudinal development of cardiovascular parameter: average heartrate | 180 days
Longitudinal development of cardiovascular parameter: maximal heartrate | 180 days
Longitudinal development of cardiovascular parameter: minimum heartrate | 180 days
Longitudinal development of cardiovascular parameter: time in light heartrate zone (seconds) Description: Light heartrate zone is defined by Withings as follows: from 0% inclusive to 50% exclusive of maximum heart rate. | 180 days
Longitudinal development of cardiovascular parameter: time in moderate heartrate zone (seconds) Description: Moderate heartrate zone is defined by Withings as follows: from 50% included to 70% excluded of maximal heart rate. | 180 days
Longitudinal development of cardiovascular parameter: time in intense heartrate zone (seconds) Description: Intense heartrate zone is defined by Withings as follows: from 70% included to 90% excluded of maximal heart rate. | 180 days
Longitudinal development of cardiovascular parameter: time in maximal heartrate zone (seconds) Description: Maximal heartrate zone is defined by Withings as follows: from 90% included to 100% included of maximal heart rate | 180 days
The Modified Ashworth Scale (MAS) | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  The Modified Ashworth Scale (MAS) is a clinical tool for assessing muscle spasticity in patients, particularly those with neurological conditions such as multiple sclerosis (MS). It assesses the resistance of a muscle to passive stretching and thus measures the degree of spasticity. The MAS helps to assess the severity of spasticity and monitor the effectiveness of treatment and disease progression. The scale ranges from 0 (no increased muscle tone) to 5 (limbs rigid in flexion and extension).

SECONDARY OUTCOMES:
WHOQoL-BREF (World Health Organization Quality of Life Questionnaire Brief Version) | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  WHOQoL-BREF (World Health Organization Quality of Life Questionnaire Brief Version): The WHOQOL-BREF questionnaire measures quality of life across 4 domains: Physical health, psychological health, social relationships and environment. It also includes one question on overall QOL and one on general health. The WHOQOL-BREF scores correlate highly (.89 or above) with WHOQOL-100 scores, and demonstrate good discriminant validity, content validity, internal consistency and test-retest reliability. The four WHOQOL-BREF domain scores will be used as main outcome measure. The measure is calculated by summing the point values for the questions corresponding to each domain and then transforming the scores to a 0-100 point interval, with higher scores corresponding to greater QOL.
The Expanded Disability Status Scale (EDSS) | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  The Expanded Disability Status Scale (EDSS) is a scale used to measure the severity of disability in patients with multiple sclerosis (MS). It assesses neurological function based on factors such as mobility, coordination, vision and strength. The scale ranges from 0 (no disability) to 10 (death due to MS). The EDSS is used to track disease progression and make treatment decisions, with higher scores indicating greater disability.
Smartwatch Questionnaire | 6 months (V3)
  Questionnaire about smartwatch usage. Patients are presented with 17 statements about the smartwatches, focusing on practicality, usability, and everyday suitability. They can score each statement from 1 to 5, where 5 means strong agreement and 1 means strong disagreement.
End of Dose Questionnaire (EOD) | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  The End-of-dose-phenomena-Questionnaire assesses the effectiveness of a treatment at the end of its dosing interval and asks about an increase in symptoms. Patients can state whether they have experienced a worsening of symptoms in recent weeks and, if so, for how many days and which migraine symptoms have worsened.
McCorkle and Young Symptom Distress Scale | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  The McCorkle and Young Symptom Distress Scale is an instrument for assessing the degree of distress caused by various physical symptoms. The scale consists of 13 symptoms (such as pain, nausea, fatigue, insomnia and shortness of breath) that are commonly experienced by patients. Patients rate each symptom on a scale of 1 to 5, with 1 being 'no distress' and 5 being 'extreme distress'. This scale can be used to determine which symptoms are the most distressing. This enables better symptom management and customised measures to improve the patient's quality of life.
The Multiple Sclerosis Impact Scale 29 (MSIS-29) | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  The Multiple Sclerosis Impact Scale 29 (MSIS-29) is a questionnaire of the impact of multiple sclerosis (MS) on patients' daily lives. It consists of 29 items divided into two sections: the physical impact (20 items) and the psychological impact (9 items) of MS. Each item is rated on a scale of 1 to 5, with a higher score indicating a greater impact. The MSIS-29 helps assess how MS affects physical function and emotional well-being and provides valuable insights for treatment planning and monitoring disease progression.
The Numeric Rating Scale (NRS) | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  The NRS is another tool used to assess pain intensity. It involves the patient rating their pain on a scale from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable." Both scales are widely used due to their simplicity and effectiveness in monitoring symptom severity.
The Montgomery-Asberg Depression Rating Scale (MADRS) | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  The Montgomery-Asberg Depression Rating Scale (MADRS) is a clinical instrument for assessing the severity of depression in patients. It consists of 10 items that assess symptoms such as mood, guilt, sleep, appetite and concentration. Each item is scored on a scale from 1 to 7, with higher scores indicating more severe depression. The MADRS is commonly used to monitor changes in depressive symptoms and evaluate the effectiveness of treatment.
The Edmonton Symptom Assessment Scale (ESAS) | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  The Edmonton Symptom Assessment Scale (ESAS) is an instrument commonly used to assess the severity of symptoms in patients with advanced or terminal illnesses. It helps to assess the intensity of symptoms such as pain, fatigue, nausea, depression, anxiety, sleep disturbance, loss of appetite, breathlessness, general well-being and physical decline. Patients rate each symptom on a scale from 0 (no symptom) to 10 (worst possible symptom), which allows for quick and effective symptom monitoring. This scale helps to adjust treatment plans and improve the quality of care by tracking changes in symptoms over time.
Sleep-Questionnaire | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  The Sleep-Questionnaire contain the Pittsburgh Sleep Quality Index (PSQI) as well as two Items on the perceived impact of the smartwatch on the patient´s sleep. The PSQI assesses the quality of sleep over a one-month interval and measures seven component scores: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Total score ranges from 0 to 21, with higher scores indicating a poorer sleep quality.
EQ-5D-5L | Screening + Baseline (V1), 3 months (V2), 6 months (V3)
  EQ-5D-5L: is a standardized instrument for measuring health-related quality of life. It assesses five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity, ranging from no problems to extreme problems. Respondents rate their health state by selecting the most appropriate level for each dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty, Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No